CLINICAL TRIAL: NCT02984943
Title: The Effects of Hyperbaric Oxygen on Rheumatoid Arthritis: A Pilot Study
Brief Title: The Effects of Hyperbaric Oxygen on Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michelle Sit, MD, Rheumatologist, David Grant U.S. Air Force Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDG20160004H
Record Dates: First submitted 2016-11-15; First posted 2016-12-07 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: RheumatoId Arthritis
Keywords: Rheumatoid Arthritis; Hyperbaric Oxygen
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hyperbaric Oxygen (Experimental): Hyperbaric Oxygen
  Interventions: Device: Hyperbaric Oxygen

INTERVENTIONS:
Device: Hyperbaric Oxygen — 30 treatments of Hyperbaric Oxygen.

SUMMARY:
The purpose of this investigation is to determine the effects and ease of using hyperbaric oxygen therapy HBO2 for the treatment of rheumatoid arthritis joint pain and prevention of disease progression. In this study it is our intention to not only evaluate effects and ease of treatment but time, cost, possible adverse events and effect size in an attempt to predict an appropriate sample size and improve on the study design prior to a more extensive study.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, systemic, inflammatory disorder of unknown etiology that primarily involves synovial joints, typically symmetrically. If untreated and/or uncontrolled, joint destruction due to erosion of cartilage and bone can cause joint destruction, joint deformities, loss of physical function, severe disability, and difficulties maintaining employment. American College of Rheumatology (ACR)/EULAR 2010 classification criteria is a score-based algorithm which adds scores of 4 categories including, joint involvement, serology, acute-phase reactants and duration of symptoms. A score of >6/10 is needed for classification of a patient as having definite RA.

Non-pharmacologic and supplementary therapies include patient education, rest, exercise, nutrition counseling, cardiovascular disease risk reduction, and immunizations to decrease risk of infectious complications of immunosuppression. These are important in the comprehensive management of RA in all stages of disease and are used in addition to drug therapy.

Pharmacologic therapies typically start with a disease-modifying anti-rheumatic drug (DMARD), preferably as soon as possible after diagnosis. DMARDs are commonly used in combination with anti-inflammatory drugs such as non-steroidal anti-inflammatory drugs (NSAIDs) and glucocorticoids which are often used as bridging therapies until the DMARDs become effective. The goal is disease remission. To assess response, disease activity scores are used along with inflammatory markers.

Three patients with active RA treated in the multi-place hyperbaric facility at David Grant Medical Center (DGMC), Travis Air Force Base, California, for non RA-related indications, all noted significant improvement in arthralgias, sleep patterns and overall well-being during the course of therapy. Two were treated at 2 atmospheres absolute (ATA) oxygen for 90 minutes daily Monday through Friday. One patient received 2 ATA air on the same treatment protocol as a participant in a research study, and a subsequent course of hyperbaric oxygen (HBO2) at 2 ATA.

This is a pilot study. Patients will be recruited through the Rheumatologists, IRB-approved HIPAA waiver to contact patients that have been seen in the military treatment facility (MTF) within the past year with a diagnosis of RA, flyers in the Rheumatology Clinic or thru Commander Calls.

During the initial screening visit:

The rheumatologist will discuss the trial and at this point the subject will be consented and the inclusion/exclusion criteria will be reviewed. If subject qualifies they will see the Hyperbaric physician who will do physical examination to determine if it is safe for the subject to receive HBO2. An human chorionic gonadotrophin (HCG) by point of care testing (POCT) will be completed by the coordinator in women capable of pregnancy. After this exam is done the subject will be scheduled for a trial Hyperbaric session.

Baseline visit will be done after the subject has tolerated the trial hyperbaric session. This visit includes:

1. A visit with the rheumatologist to do routine assessments to establish baseline measurement using the Disease Activity Scale (DAS28)
2. Labs (CRP and Erythrocyte Sedimentation Rate (ESR), basic metabolic panel (BMP) and microparticles), will be completed. Magnetic resonance imaging (MRI) with and without contrast and ultrasound will be done on both hands from wrists to proximal phalanges the wrist. BMP is done pre-MRI to guarantee adequate kidney function.
3. Subjective patient reporting will be captured using the Routine Assessment of Patient Index Data (RAPID 3)
4. Sleep quality will be tracked using the Pain and Sleep Quality Questionnaire (PSQ-3).
5. Visual Analog Scores (VAS) for pain will be tracked.
6. Surveys will be done by a study team member

The subject at this time will be scheduled to start HBO2 treatments. Screening, baseline, first HBO2 treatment all in one month. Participants will complete 30 sessions within 10 weeks.

If the subject reports pain relief (> 40% or zero pain) during the HBO2 treatments the will be referred to the rheumatologist for assessment. Pain improvement will be based on a pain assessment (1-10 scale reported verbally) at hyperbaric treatment visits. Labs will be drawn at this time. RAPID 3, PSQ-3 and VAS will be done at least six times while undergoing HBO2 treatment to track subject progress. Labs (CRP, ESR, microparticles) will be repeated at the conclusion of the HBO2 treatments.

At the month 3 and month 6 visit (+/- 2 week window) the subject will see the rheumatologist to track disease activity using the DAS-28. The date of the visit will be scheduled for three and six months from the baseline visit. The rheumatologist will order the MRI, ultrasound and lab studies prior to the visit. RAPID 3, PSQ-3 and VAS will be administered at this time. Lab samples will be collected prior to the Rheumatology appointment.

The six month visit marks the end of the trial. Patients will continue to be followed in Rheumatology Clinic every three months.

If the patient's RA symptoms worsen during the study, the physicians will institute measures to address the cause. The medical monitor will be notified and if any adverse events are involved, they will be recorded and reported to the Institutional Review Board (IRB).

Data:

Data will be entered by authorized study personnel only. Demographic information will be collected including sex, age and ethnic background in accordance with HIPPA compliance.

Data collected during this study will be analyzed at various points in time to include physician exams, labs (CRP, ESR, BMP, analysis of microparticles, neutrophil and platelet activation), radiologic studies, joint inspection.

Changes in joint pain will be determined by self-reporting and results of the standard outcome measures questionnaires (RAPID 3, PSQ-3 and VAS). A separate sleep survey will be administered.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Active duty or Department of Defense (DoD) beneficiary
3. Diagnosed with rheumatoid arthritis meeting ACR/EULAR 2010 classification criteria and any one of the following:

   1. Patient does not want to be on rheumatologic medications
   2. Patient has contraindications to standard rheumatologic medications
   3. Patient has failed treatment or an incomplete response with standard rheumatologic medications
4. Women of childbearing age must have a negative pregnancy test and currently be on a reliable form of birth control

Exclusion Criteria:

1. Severe depression
2. Dementia, mental disability
3. Claustrophobia
4. Uncontrolled seizure disorder
5. Uncontrolled asthma/severe chronic obstructive pulmonary disease (COPD) with partial pressure of carbon dioxide (pCO2) > 45 mmHg on arterial blood gas
6. Grade 4 congestive heart failure
7. Unstable angina
8. Chronic/acute otitis media/sinusitis
9. Major tympanic membrane trauma
10. Severe kyphoscoliosis
11. Prior chemotherapy with Bleomycin and evidence of deterioration in diffusion capacity of the lung for carbon monoxide (DLCO) after a single hyperbaric oxygen exposure
12. History of renal insufficiency or glomerular filtration rate (GFR)< 30
13. Women that are currently pregnant or breast feeding or intend on becoming pregnant while enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle T Sit, MD, Principal Investigator — David Grant Medical Center. Travis AFB
Locations (1):
- David Grant Medical Center, Travis Air Force Base, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Ann Rheum Dis. 2010 Sep;69(9):1580-8. doi: 10.1136/ard.2010.138461. PMID 20699241
- [Background] Ayearst L, Harsanyi Z, Michalko KJ. The Pain and Sleep Questionnaire three-item index (PSQ-3): a reliable and valid measure of the impact of pain on sleep in chronic nonmalignant pain of various etiologies. Pain Res Manag. 2012 Jul-Aug;17(4):281-90. doi: 10.1155/2012/635967. PMID 22891194
- [Background] Pincus T, Swearingen C, Wolfe F. Toward a multidimensional Health Assessment Questionnaire (MDHAQ): assessment of advanced activities of daily living and psychological status in the patient-friendly health assessment questionnaire format. Arthritis Rheum. 1999 Oct;42(10):2220-30. doi: 10.1002/1529-0131(199910)42:103.0.CO;2-5. PMID 10524697
- [Result] Varga OIu, Ignat'ev VK, Vezikova NN, Kheifetz IV. [Radiation-modifying effect of oxygen barotherapy in complex treatment of patients with rheumatoid arthritis and osteoarthrosis]. Ter Arkh. 2002;74(12):83-6. Russian. PMID 12577851
- [Derived] Sit MT, Schmidt TW, Edmonds LD, Kelly JA, Sky KM, Thornton JA, McNeary-Garvin AM, Thom SR, Slade JB. The Effects of Hyperbaric Oxygen on Rheumatoid Arthritis: A Pilot Study. J Clin Rheumatol. 2021 Dec 1;27(8):e462-e468. doi: 10.1097/RHU.0000000000001540. PMID 32947434
- See also: Hyperbaric oxygen in chronic traumatic brain injury: oxygen, pressure, and gene therapy — http://www.medicalgasresearch.com/conten/5/1/9
- See also: Disease activity score for rheumatoid arthritis. — http://www.das-score.nl
- See also: Approaches to the management of rheumatoid arthritis — https://www.uptodate.com/contents/assessment-of-rheumatoid-arthritis-activity-in-clinical-trials-and-clinical-practice?source=search_result&search=assessment%20of%20reumatoid%20arthritis%20activity%20in%20clinical%20trial%20and%20clinical%20practive&selectedTitle=2~150
- See also: The treatment of rheumatoid arthritis (RA) is directed toward the control of synovitis and the prevention of joint injury. — https://www.uptodate.com/contents/general-principles-of-management-of-rheumatoid-arthritis-in-adults?source=search_result&search=general%20principles%20of%20management%20of%20rheumatoid%20arthritis%20in%20adults&selectedTitle=1~150

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyperbaric Oxygen
Started | 14
Completed | 10
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: A total of 14 participants were enrolled. 3 participants withdrew. 1 physician decision
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
Age, Customized [Mean (Standard Deviation); unit: years] — Population: 3 participant withdrew
  1 physician decision
  years
    Age >/= 18 | 66.3 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 participant withdrew
  1 physician decision
  Participants
    Female | 7
    Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 3 participants withdrew
  1 physician decision
  Participants
    Caucasian | 6
    Asian | 4
    Native American | 0
    Hispanic | 0
Diagnosed with rheumatoid arthritis meeting ACR/EULAR 2010 classification and 1 other criteria [Count of Participants; unit: Participants] — additional criteria (at least one)
  1. Patient does not want to be on rheumatologic medications.
  2. Patient has contraindications to standard rheumatologic medications.
  3. Patient has failed treatment or an incomplete response with standard rheumatologic medications. Population: 3 participants withdrew
  1 physician decision
  Participants | 10

OUTCOME MEASURES:

1. Primary Outcome: Sleep Quality - Trouble Falling Asleep, 6 Weeks
Description: The Pain Sleep Quality (PSQ)-3 questionnaire will be used to measure outcome. Participants will score the question "How often have you had trouble falling asleep because of pain?" by placing a slash (/) on a 10 cm line directly beneath the question. The line will have "never" and "always" at each end. A ruler will be used to determine were the slash falls. The value between, 0-10, that corresponds on the ruler with the slash will be documented. "0" is a better outcome, and "10" is a worse outcome. The value for each participant will be combined to obtain a median and inter-quartile range at 6 weeks
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 1.3 [0.5 to 2.4]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.10, Skillings-Mack test

2. Primary Outcome: Sleep Quality - Trouble Falling Asleep, 6 Months
Description: The PSQ-3 questionnaire will be used to measure outcome. Participants will score the question "How often have you had trouble falling asleep because of pain?" by placing a slash (/) on a 10 cm line directly beneath the question. The line will have "never" and "always" at each end. A ruler will be used to determine were the slash falls. The value between, 0-10, that corresponds on the ruler with the slash will be documented. "0"is a better outcome, and "10" is a worse outcome. The value for each participant will be combined to report a median and inter-quartile range at 6 months.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 0.9 [0.5 to 3.5]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.10, Skillings-Mack test

3. Primary Outcome: Sleep Quality - Morning Pain, 6 Weeks
Description: The PSQ-3 questionnaire will be used to measure outcome. Participants will score the question "How often have you been awakened by pain during the morning?" by placing a slash (/) on a 10 cm line directly beneath the question. The line will have "never" and "always" at each end. A ruler will be used to determine were the slash falls. The value between, 0-10, that corresponds on the ruler with the slash will be documented. "0"is a better outcome, and "10" is a worse outcome. The value for each participant will be combined to report a median and inter-quartile range at 6 weeks
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 1.1 [0.3 to 1.5]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.02, Skillings-Mack test

4. Primary Outcome: Sleep Quality - Morning Pain, 6 Months
Description: The PSQ-3 questionnaire will be used to measure outcome. Participants will score the question "How often have you been awakened by pain during the morning?" by placing a slash (/) on a 10 cm line directly beneath the question. The line will have "never" and "always" at each end. A ruler will be used to determine were the slash falls. The value between, 0-10, that corresponds on the ruler with the slash will be documented. "0"is a better outcome, and "10" is a worse outcome. The value for each participant will be combined to report a median and inter-quartile range at 6 months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 0.8 [0 to 5.2]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.02, Skillings-Mack test

5. Primary Outcome: Sleep Quality - Night Pain, 6 Weeks
Description: The PSQ-3 questionnaire will be used to measure outcome. Participants will score the question "How often have you been awakened by pain during the night?" by placing a slash (/) on a 10 cm line directly beneath the question. The line will have "never" and "always" at each end. A ruler will be used to determine were the slash falls. The value between, 0-10, that corresponds on the ruler with the slash will be documented. "0"is a better outcome, and "10" is a worse outcome. The value for each participant will be combined to report a median and inter-quartile range at 6 weeks
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 1.1 [0.5 to 2.5]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.004, Skillings-Mack test

6. Primary Outcome: Sleep Quality - Night Pain, 6 Months
Description: The PSQ-3 questionnaire will be used to measure outcome. Participants will score the question "How often have you been awakened by pain during the night?" by placing a slash (/) on a 10 cm line directly beneath the question. The line will have "never" and "always" at each end. A ruler will be used to determine were the slash falls. The value between, 0-10, that corresponds on the ruler with the slash will be documented. "0"is a better outcome, and "10" is a worse outcome. The value for each participant will be combined to report a median and inter-quartile range at 6 months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 1.2 [0 to 4]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.004, Skillings-Mack test

7. Primary Outcome: DAS28 - Global Health (GH), 3 Months
Description: DAS28 quantifies disease activity based on visual analogue scales (VAS) assessment of well-being rated on a scale of 0-100 mm."0"is a better outcome, and "100" is a worse outcome. The value for each participant will be combined to obtain a median and inter-quartile range at 3 months
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 30 [15 to 50]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.2938, Skillings-Mack test

8. Primary Outcome: DAS28 - Global Health (GH), 6 Months
Description: DAS28 quantifies disease activity based on visual analogue scales (VAS) assessment of well-being rated on a scale of 0-100 mm. "0"is a better outcome, and "100" is a worse outcome. The value for each participant will be combined to obtain a median and inter-quartile range at 6 months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 30 [10 to 50]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.2938, Skillings-Mack test

9. Primary Outcome: DAS28 - C-reactive Protein (CRP), 3 Months
Description: DAS28 quantifies disease activity based on a mathematical formula that computes four variables: number of swollen and tender joints (total number of joints assessed is 28), CRP (mg/L) and visual analogue scales (VAS) for patient global assessment of well-being (0-100 mm). "0"is a better outcome, and "100" is a worse outcome. The value for each participant will be combined to obtain a median and inter-quartile range at 3 months
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 3.1 [2.3 to 4.0]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.0608, Skillings-Mack test

10. Primary Outcome: DAS28 - C-reactive Protein (CRP), 6 Months
Description: DAS28 quantifies disease activity based on a mathematical formula that computes four variables: number of swollen and tender joints (total number of joints assessed is 28), CRP (mg/L) and visual analogue scales (VAS) for patient global assessment of wellbeing (0-100 mm). "0"is a better outcome, and "100" is a worse outcome. The value for each participant will be combined to obtain a median and inter-quartile range at 6 months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 3.1 [2.2 to 3.8]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.0608, Skillings-Mack test

11. Primary Outcome: DAS28 - Erythrocyte Sedimentation Rate (ESR), 3 Months
Description: DAS28 quantifies disease activity based on a mathematical formula that computes four variables: number of swollen and tender joints (total number of joints assessed is 28), ESR (mm/h) and visual analogue scales (VAS) for patient global assessment of well-being (0-100 mm). "0"is a better outcome, and "100" is a worse outcome. The value for each participant will be combined to obtain a median and inter-quartile range at 3 months
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 4.1 [2.3 to 4.8]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.1496, Skillings-Mack test

12. Primary Outcome: DAS28 - Erythrocyte Sedimentation Rate (ESR), 6 Months
Description: DAS28 quantifies disease activity based on a mathematical formula that computes four variables: number of swollen and tender joints (total number of joints assessed is 28), ESR (mm/h) and visual analogue scales (VAS) for patient global assessment of well-being (0-100 mm). "0"is a better outcome, and "100" is a worse outcome. The value for each participant will be combined to obtain a median and inter-quartile range at 6 months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 3.8 [3.0 to 3.9]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.1496, Skillings-Mack test

13. Primary Outcome: RAPID 3 - Abilities, 6 Weeks
Description: A questionnaire that assesses abilities on a scale of 0-10. "0"is a better outcome, and "10" is a worse outcome. The value for each participant will be combined to report a median and inter-quartile range at 6 weeks.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 1.5 [0.0 to 2.7]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.36, Skillings-Mack test

14. Primary Outcome: RAPID 3 - Abilities, 6 Months
Description: A questionnaire that assesses abilities on a scale of 0-10. "0"is a better outcome, and "10" is a worse outcome. The value for each participant will be combined to report a median and inter-quartile range at 6 months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 1.9 [0.7 to 2.3]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.36, Skillings-Mack test

15. Primary Outcome: RAPID 3 - Pain, 6 Weeks
Description: A questionnaire that assesses pain on a scale of 0-10. "0"is a better outcome, and "10" is a worse outcome. The value for each participant will be combined to report a median and inter-quartile range at 6 weeks
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 2.5 [0.5 to 3.5]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.0012, Skillings-Mack test

16. Primary Outcome: RAPID 3 - Pain, 6 Months
Description: A questionnaire that assesses pain on a scale of 0-10. "0"is a better outcome, and "10" is a worse outcome. The value for each participant will be combined to report a median and inter-quartile range at 6 months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 2.3 [0.5 to 4.5]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.0012, Skillings-Mack test

17. Primary Outcome: RAPID 3 - Illness/Health, 6 Weeks
Description: A questionnaire that assesses illness/health on a scale of 0-10. "0"is a better outcome, and "10" is a worse outcome. The value for each participant will be combined to report a median and inter-quartile range at 6 weeks
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 3.3 [0.5 to 5.0]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.90, Skillings-Mack test

18. Primary Outcome: RAPID 3 - Illness/Health, 6 Months
Description: A questionnaire that assesses illness/health on a scale of 0-10. "0"is a better outcome, and "10" is a worse outcome. The value for each participant will be combined to report a median and inter-quartile range at 6 months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 3.5 [1.0 to 4.5]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.90, Skillings-Mack test

19. Primary Outcome: RAPID 3 - Cumulative Scores, 6 Weeks
Description: The combined abilities, pain and illness/health scores. Recorded as a number between 0-30. "0"is a better outcome, and "30" is a worse outcome. The value for each participant will be combined to report a median and inter-quartile range at 6 weeks
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 8.4 [2.7 to 9.8]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.0068, Skillings-Mack test

20. Primary Outcome: RAPID 3 - Cumulative Scores, 6 Months
Description: The combined abilities, pain and illness/health scores. Recorded as a number between 0-30. "0"is a better outcome, and "30" is a worse outcome. The value for each participant will be combined to report a median and inter-quartile range at 6 months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 8.5 [2.0 to 12.2]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.0068, Skillings-Mack test

21. Primary Outcome: RAPID 3 - Weighed Scores, 6 Weeks
Description: The cumulative score conversion (based on a table). Recorded as a number between 0-10. 0-1 is near remission, 1.3-2 is low severity, 2.3 -4 is moderate severity, and 4.3 - 10 is high severity. The value for each participant will be combined to report a median and inter-quartile range at 6 weeks
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 2.9 [1.0 to 3.3]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.0183, Skillings-Mack test

22. Primary Outcome: RAPID 3 - Weighed Scores, 6 Months
Description: The cumulative score conversion (based on a table). Recorded as a number between 0-10. 0-1 is near remission, 1.3-2 is low severity, 2.3 -4 is moderate severity, and 4.3 - 10 is high severity. The value for each participant will be combined to report a median and inter-quartile range at 6 months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 2.7 [0.7 to 4.0]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.0183, Skillings-Mack test

23. Primary Outcome: VAS Pain Scale - 6 Weeks
Description: A pain assessment using a horizontal line with numbers, 0-10, along the axis with endpoints "no pain" to "worse possible pain". "0"is a better outcome, and "10" is a worse outcome. Participants will mark on the line the level of pain they are experiencing now. The value for each participant will be combined to report a median and inter-quartile range at 6 weeks
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 2.1 [0.825 to 2.925]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.08, Skillings-Mack test

24. Primary Outcome: VAS Pain Scale - 6 Months
Description: A pain assessment using a horizontal line with numbers, 0-10, along the axis with endpoints "no pain" to "worse possible pain". "0"is a better outcome, and "10" is a worse outcome. Participants will mark on the line the level of pain they are experiencing now. The value for each participant will be combined to report a median and inter-quartile range at 6 months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 10
score on a scale | 2.5 [0.625 to 3.5]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; p = 0.08, Skillings-Mack test

25. Primary Outcome: MRI - Synovitis, Combined Score (CS), Right, 3 Months
Description: Each of the 23 joints in the hand/wrist will be assigned a score from 0-3 based on the proportion of bone involved. "0" is best outcome, "3"worse outcome. The median score of all 23 joints at baseline and 3 months will then be calculated for each participant. Participants with a lower median score at 3 months relative to baseline will be considered "improved" for the 3 month time point. The number of participants with "improved" scores will be added to form the total number with improvement at 3 months
Time Frame: 3 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 1
  Without Improvement | 8
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; Descriptive statistics only were used

26. Primary Outcome: MRI - Synovitis, Combined Score (CS), Right, 6 Months
Description: Each of the 23 joints in the hand/wrist will be assigned a score from 0-3 based on the proportion of bone involved. "0" is best outcome, "3"worse outcome. The median score of all 23 joints at baseline and 6 months will then be calculated for each participant. Participants with a lower median score at 6 months relative to baseline will be considered "improved" for the 6 month time point. The number of participants with "improved" scores will be added to form the total number with improvement at 6 months
Time Frame: 6 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 0
  Without Improvement | 9
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; Descriptive statistics only were used

27. Primary Outcome: MRI - Synovitis, Combined Score (CS), Left, 3 Months
Description: as for outcome 25
Time Frame: 3 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 1
  Without Improvement | 8
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; Descriptive statistics only were used

28. Primary Outcome: MRI - Synovitis, Combined Score (CS), Left, 6 Months
Description: as for outcome 26
Time Frame: 6 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 2
  Without Improvement | 7
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; Descriptive statistics only were used

29. Primary Outcome: MRI - Bone Erosion, Combined Score (CS), Right, 3 Months
Description: Each of the 23 joints in the hand/wrist will be assigned a score from 0-10 based on the proportion of bone involved. "0" is best outcome, "10"worse outcome. The median score of all 23 joints at baseline and 3 months will then be calculated for each participant. Participants with a higher median score at 3 months relative to baseline will be considered "improved" for the 3 month time point. The number of participants with "improved" scores will be added to form the total number with improvement at 3 months
Time Frame: 3 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 9
  Without Improvement | 0
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; Descriptive statistics only were used

30. Primary Outcome: MRI - Bone Erosion, Combined Score (CS), Right, 6 Months
Description: Each of the 23 joints in the hand/wrist will be assigned a score from 0-10 based on the proportion of bone involved. "0" is best outcome, "10"worse outcome. The median score of all 23 joints at baseline and 6 months will then be calculated for each participant. Participants with a higher median score at 6 months relative to baseline will be considered "improved" for the 6 month time point. The number of participants with "improved" scores will be added to form the total number with improvement at 6 months
Time Frame: 6 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 9
  Without Improvement | 0
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; Descriptive statistics only were used

31. Primary Outcome: MRI - Bone Erosion, Combined Score (CS), Left, 3 Months
Description: as for outcome 29
Time Frame: 3 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 9
  Without Improvement | 0
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; Descriptive statistics only were used

32. Primary Outcome: MRI - Bone Erosion, Combined Score (CS), Left, 6 Months
Description: as for outcome 30
Time Frame: 6 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 9
  Without Improvement | 0

33. Primary Outcome: MRI - Oedema, Combined Score (CS), Left, 3 Months
Description: as for outcome 25
Time Frame: 3 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 1
  Without Improvement | 8
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; Descriptive statistics only were used

34. Primary Outcome: MRI - Oedema, Combined Score (CS), Left, 6 Months
Description: as for outcome 26
Time Frame: 6 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 1
  Without Improvement | 8
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; Descriptive statistics only were used

35. Primary Outcome: MRI - Oedema, Combined Score (CS), Right, 3 Months
Description: as for outcome 25
Time Frame: 3 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 0
  Without Improvement | 9
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; Descriptive statistics only were used

36. Primary Outcome: MRI - Oedema, Combined Score (CS), Right, 6 Months
Description: as for outcome 26
Time Frame: 6 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 0
  Without Improvement | 9

37. Primary Outcome: Ultrasound - Synovitis, Combined Score (CS), Right, 3 Months
Description: as for outcome 25
Time Frame: 3 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 1
  Without Improvement | 8
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; Descriptive statistics only were used

38. Primary Outcome: Ultrasound - Synovitis, Combined Scale (CS), Right - 6 Months
Description: as for outcome 26
Time Frame: 6 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 1
  Without Improvement | 8
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; Descriptive statistics only were used

39. Primary Outcome: Ultrasound - Synovitis, Combined Score (CS), Left, 3 Months
Description: as for outcome 25
Time Frame: 3 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 1
  Without Improvement | 8
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; Descriptive statistics only were used

40. Primary Outcome: Ultrasound - Synovitis, Combined Score (CS), Left, 6 Months
Description: Each of the 23 joints in the hand/wrist will be assigned a score from 0-3 based on the proportion of bone involved. "0" is best outcome, "3"worse outcome. The median score of all 23 joints at baseline and 6 months will then be calculated for each participant. Participants with a lower median score at 6 months relative to baseline will be considered "improved" for the t month time point. The number of participants with "improved" scores will be added to form the total number with improvement at t months
Time Frame: 6 months
Population: 10 participants imaged. 1 unable to analyze due to fusion on imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen
Number analyzed (Participants) | 9
Participants
  Improvement | 1
  Without Improvement | 8
Statistical Analysis 1: Comparison: Hyperbaric Oxygen; Test type: Other; Descriptive statistics only were used

ADVERSE EVENTS:
Time Frame: through study completion, an average of 6 months
Arm/Group | Hyperbaric Oxygen
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperbaric Oxygen (N=10)
Diffuse pruritus & popular rash (Skin and subcutaneous tissue disorders) | 1 (1) — Onset of symptoms following carpal tunnel surgery, 26 Jul 18
Left knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Diagnosed as ilio-tibial band syndrome associated with activity
Interstitial Lung Disease (ILD) (Respiratory, thoracic and mediastinal disorders) | 1 (1) — ILD is a condition associated with Rheumatoid Arthritis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT02984943/Prot_SAP_000.pdf